CLINICAL TRIAL: NCT01215214
Title: Identification and Evaluation of Endogenous Markers for the Assessment of CYP3A Activity Using Metabolomics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Education Science and Technology, Korea (Other)
Responsible Party: Joo-Youn Cho, Seoul National University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SNUCPT10_CYP3A
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: metabolite profiles; pharmacokinetics; CYP3A; metabolomics
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- midazolam (Experimental): period 1: midazolam administration alone period 2: ketoconazole 400 mg PO for 4 days administration, midazolam iv single administration period 3: rifampicin 600 mg PO for 9 days administration, midazolam iv single administration
  Interventions: Drug: midazolam

INTERVENTIONS:
Drug: midazolam — midazolam: 3mg iv
  Other Names: Bukwang midazolam, Korea

SUMMARY:
Identification and evaluation of endogenous markers for the assessment of CYP3A activity using metabolomics.

DETAILED DESCRIPTION:
Eligibility for participation of this study will be determined from demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 3 weeks before study drug administration. Subjects suitable for this study will be admitted to the Clinical Trials Center, Seoul National University Hospital on the day before dosing, and they were overnight-fasted from 10 p.m. of Day -1. Urine collection is scheduled drug 24 hour before midazolam administration. Subjects will be dosed study drug via intravenous around at 9 a.m. of Day 1. Subjects performed scheduled procedures including clinical laboratory tests, electrocardiograms and pharmacokinetic samplings. Subjects will be discharged on Day 2, and visited Clinical Trials Center on Day 5-7 for ketoconazole administration. Subjects will be admitted on Day 7 for period 2. Subjects performed scheduled period 2 (ketoconazole co-administration phase), and period 3 (rifampicin co-administration phase) procedure. Study participation was terminated on post-study visit (Day 30-32).

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20 to 50 years of age, inclusive
* Weight: Between 50 - 95 kg, within 17-28 of Body Mass Index
* Subject who are reliable and willing to make themselves available during the study period, are willing to follow the study protocol, and give their written informed consent voluntarily

Exclusion Criteria:

* History of hypersensitive reaction to medication (midazolam, ketoconazole, rifampicin)
* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease History or evidence of drug abuse
* Use any prescriptive medication, Korean traditional medication not considered acceptable by the clinical investigator during the last 14 days period before first dosing, or use any OTC medication not considered acceptable by the clinical investigator during the last 7 days period before first dosing (if used medication is considered acceptable by investigator, patients can be included)
* Participation in clinical trials of any drug within 60 days prior to the participation of the study
* Judged to be inappropriate for the study by the investigator

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Metabolomic profile | -24- -12h, -12- 0h of every midazolam dosing
  endogenous metabolite profiles such as steroids

SECONDARY OUTCOMES:
Pharmacokinetics | 0h, 10m, 20m, 30m, 45m, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h
  Cmax, AUClast of midazolam

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Youn Cho, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea